CLINICAL TRIAL: NCT05946161
Title: A Digital Intervention Program to Promote Mental and Sexual Health of Prostate Cancer Survivors
Brief Title: Testing an e-Health Intervention for Prostate Cancer Survivors' Mental and Sexual Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Collaborators: Horizon 2020 - European Commission (Other)
Responsible Party: Principal Investigator, Ana Luísa de Matos Dias Quinta Gomes, Assistant Researcher, Universidade do Porto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NORTE-01-0145-FEDER-000057
Record Dates: First submitted 2023-06-23; First posted 2023-07-14 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Prostate Cancer
Keywords: e-Health; cognitive behavioral therapy; prostate cancer; sexual health; mental health
MeSH Terms: conditions — Prostatic Neoplasms; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- testing the digital intervention (Experimental): Prostate cancer survivors (n=20) randomly assigned to this arm will complete a digital psychosexual intervention and will be accompanied weekly by a certified clinical psychologist to monitor progress (synchronous or asynchronous). Pre and Post testing involve questionnaires collecting data on psychosexual variables. At post-testing a 30-minute interview will be conducted to collect information on the usability
  Interventions: Behavioral: e-Health intervention to promote mental and sexual health of prostate cancer survivors
- waiting list (No Intervention): Prostate cancer survivors (n=20) randomly assigned to this arm will not be accompanied or get access to the intervention during the six week period in which the experimental group is completing the intervention. Pre and Post testing involved questionnaires collecting data on psychosexual variables. After post testing the control arm will gain access to the intervention as compensation for their participation

INTERVENTIONS:
Behavioral: e-Health intervention to promote mental and sexual health of prostate cancer survivors — An online psychological intervention (e-Health app technology) specifically tailored to meet the needs of Portuguese men with prostate cancer was developed to promote participants' mental and sexual health. The intervention protocol was designed under the principles of Cognitive Behavior Therapy (CBT), featuring psychological and sexual health promotion strategies. The intervention program consists of 5 modules covering components of psychoeducation, sexual rehabilitation, mindfulness, cognitive restructuring and relapse prevention. The modules will be delivered online (using text, videos, and graphics) along with therapeutic guidance and support provided by a certified Clinical Psychologist, over a 6-week period.
  Arms: testing the digital intervention

SUMMARY:
This study aims to assess the acceptability, feasibility, and preliminary efficacy of an e-Health psychological intervention specifically designed to promote sexual health, mental health, and general well-being and quality of life in men with prostate cancer. A pilot study will be conducted involving prostate cancer survivors randomly assigned to one of two conditions: the experimental group (receiving the program) vs the control condition (waiting list). The experimental group is expected to improve on outcomes related to mental and sexual well-being when compared to the control group. Furthermore, the experimental group is expected to show good acceptability of the intervention program. This study aims to inform the design and methodology to be adopted in a future randomized controlled trial aimed to further test the e-Health intervention's efficacy.

DETAILED DESCRIPTION:
This study was approved by the Ethical Board of São João Hospital, Porto. An online psychological intervention (e-Health app technology) specifically tailored to meet the needs of Portuguese men with prostate cancer was developed to promote participants' mental and sexual health. The intervention protocol was designed under Cognitive-Behavior Therapy (CBT) principles, featuring psychological and sexual health promotion strategies. The intervention program consists of 5 modules covering components of psychoeducation, sexual rehabilitation, mindfulness, cognitive restructuring, and relapse prevention. The modules will be delivered online (using text, videos, and graphics) along with therapeutic guidance and support provided by a certified Clinical Psychologist over six weeks.

Participants will be recruited at cancer units and will meet the inclusion criteria: prostate cancer survivors; 18 years old or older; ability to give informed consent; regular use of a smartphone and internet access; no other oncological diagnoses over the past five years, no severe neurological or psychological disorders. Participants will be randomly assigned to one of two conditions: 1) e-Health psychological intervention (N = 20); 2) waiting list group, N = 20). Participants will be clinically assessed before and after intervention on different psychosexual dimensions (e.g., mental health, quality of life, sexual dysfunction). By the end of the study, the waiting list group participants will be allowed to access the e-Health psychological intervention. The experimental group is expected to improve regarding mental and sexual well-being outcomes compared to the control group. Furthermore, the experimental group is expected to show the program's acceptability. This study aims to inform a future a randomized control trial that aims to further test the e-Health intervention's efficacy. Pre, post-test, and 3-month follow-up assessments will be performed.

Main outcomes: psychological distress, sexual distress, sexual satisfaction, relational satisfaction, sexual dysfunctional beliefs, and quality of life. All scales are validated and adapted to the Portuguese population. Furthermore, a semi-structured interview will be conducted with experimental group participants by the end of the study to collect user feedback.

Participants' data will be stored in an encrypted file, saved on a computer, and only accessible to the main researchers of this study. Confidentiality will be guaranteed by attributing an individual code to each participant. This code will be used to log into the digital intervention and complete psychometric scales. Interviews will be recorded and transcribed. Transcriptions will be marked with the same code to ensure the association of the collected data.

Statistical procedures will be performed using IBM SPSS and include i) descriptive analyses; ii) MANOVA to measure differences among groups and to compare assessment moments; iii) thematic analysis to understand the user's experience (post-intervention interview)

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer survivors,
* 18 years old or older,
* Ability to give informed consent,
* Regular use of a smartphone and internet access.

Exclusion Criteria:

* Other diagnosed oncological diseases over the past five years,
* Severe neurological impairment or other severe psychological/psychiatric diseases (depression, generalized anxiety disorder, psychosis-related disorders),
* Other uncontrolled/unstable diseases,
* Severe hearing and/or visual impairment,
* Under psychotherapy or treatment for sexual problems,
* Participating concurrently in other clinical trials.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Brief Symptom Inventory | Change from baseline psychological distress at final program (6 weeks)
  Questionnaire to assess psychological distress
Sexual Distress Scale | Change from baseline sexual distress at final program (6 weeks)
  Questionnaire to assess sexual distress
WHOQoL-BREF | Change from baseline quality of life at final program (6 weeks)
  Questionnaire to assess quality of life
Global Measure of Sexual Satisfaction | Change from baseline sexual satisfaction at final program (6 weeks)
  Questionnaire to assess sexual satisfaction
Global Measure of Relationship Satisfaction | Change from baseline relationship satisfaction at final program (6 weeks)
  Questionnaire to assess relationship satisfaction
System Usability Scale | Post assessment - through study completation, (6 weeks)
  Questionnaire to assess acceptability and usability

SECONDARY OUTCOMES:
International Index of Erectile Function | Change from baseline sexual function at final program (6 weeks)
  Questionnaire to assess sexual function
Dysfunctional Sexual Beliefs Questionnaire | Change from baseline dysfunctional sexual beliefs at final program (6 weeks)
  Questionnaire to assess dysfunctional sexual beliefs

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Psychology and Educational Sciences, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No